CLINICAL TRIAL: NCT06758141
Title: Using 3D Printed Advanced Cardiac Models for Transseptal Puncture, Cardiac Ablation, and Cardiac Tamponade Simulation Training to Enhance Medical Education: a Randomized Controlled Educational Trial
Brief Title: 3D Printed Advanced Cardiac Models for Transseptal Puncture, Cardiac Ablation, and Cardiac Tamponade Simulation Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Assistant Professor, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FJUH113381
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Satisfaction, Personal
Keywords: clinical simulation-based education; advanced cardiology procedures; transseptal puncture; cardiac ablation; cardiac tamponade
MeSH Terms: conditions — Personal Satisfaction; Cardiac Tamponade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D-printed presention group (Experimental): Received a routine presentation plus 3D printing model
  Interventions: Other: 3D printed educational model
- Slide-based presention group (Active Comparator): Received a routine presentation
  Interventions: Other: Slide-based presentation

INTERVENTIONS:
Other: 3D printed educational model — 3D Printed Advanced Cardiac Model
  Arms: 3D-printed presention group
Other: Slide-based presentation — Slide-based presentation
  Arms: Slide-based presention group

SUMMARY:
The objective of this study is to develop advanced cardiac models using 3D printing technology for teaching complex cardiology procedures such as (1) transseptal puncture, (2) cardiac ablation, and (3) ultrasound scanning and drainage of cardiac tamponade. By implementing this study, the investigators aim to transform the teaching methods for cardiology students at our hospital.

DETAILED DESCRIPTION:
Background： The standard methodology for education in medicine, particularly in cardiology, still follows the apprenticeship model, where trainees observe, gradually take over, and practice under supervision until they can independently perform procedures. The traditional pedagogical strategy for complex medical procedures, like cardiac catheterization, emphasizes the "see one, do one, teach one" doctrine. Studies have revealed the superior efficacy of 3D printing in medical education, particularly in enhancing learning skills and knowledge among medical students. The demand for 3D printed models in medical education is increasing continuously.

Study Design：

This study is a single-center, pilot, prospective, randomized controlled educational trial.

Methods：

The trial will be conducted in the Department of Cardiovascular Medicine at Fu Jen Catholic University Hospital. The investigators plan to enroll 50 participants, who will be randomly assigned to either the 3D model training group (n=25) or the conventional curriculum group (n=25) in a 1:1 ratio. All participants will undergo pre- and post-training assessments, including a knowledge test (structured written questionnaire), an attitude assessment (semi-structured satisfaction questionnaire), and a skills evaluation (direct observation of procedural skills, DOPS).

Effect：

The investigators anticipate the development of a set of advanced 3D cardiac models for teaching cardiology procedures. It is expected that combining classroom learning with the viewing and interactive practice of 3D printed models will significantly improve the learning outcomes of the trainees.

Key words：

Clinical simulation-based education, advanced cardiology procedures, transseptal puncture, cardiac ablation, cardiac tamponade.

ELIGIBILITY:
Inclusion Criteria:

* Medical student, nurse practitioner and Resident in Fu Jen Catholic University Hospital

Exclusion Criteria:

* Refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Examination score of pre-intervention | pre-intervention
  score of pre-intervention (maximun 100 and minimum 0), higher means a better outcome
Examination score of post-intervention | immediately after the intervention
  score of post-intervention (maximun 100 and minimum 0), higher means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No